CLINICAL TRIAL: NCT03930134
Title: Sparse Uterine Closure in Caesarean Section: Short and Mid Term Results
Brief Title: Sparse Uterine Closure in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaouther Dimassi, associate professor in obstetrics and gynecology, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: sparse uterine closure
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Caesarean Scar Defect
Keywords: caesarean; scar defect; sparse uterine suture; one layer uterine suture; blood loss; ultrasound
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sparse uterine suture (Experimental): women who had a french ambulatory casarean section including a sparse uterine closure
  Interventions: Procedure: sparse uterine suture
- one layer uterine closure (Active Comparator): women who had a misgav ladach caesarean section section, including a one layer classical uterine closure
  Interventions: Procedure: one layer uterine closure

INTERVENTIONS:
Procedure: sparse uterine suture — The slowly absorbed Vicryl 1 suture with a large round needle is introduced intramyometrially right above the endometrium. The suture starts in one corner and proceeds along the lower then the upper edge returning back to the incision point. Subserous layer is closed upon using the same thread in order to cover the purse suture and to complete the haemostasis while increasing the wound thickness.
  Arms: sparse uterine suture
Procedure: one layer uterine closure — one layer classical continious uterine closure using slowly absorbed Vicryl 1
  Arms: one layer uterine closure

SUMMARY:
The existence and the characteristics of a wedge- shaped defect in the uterine incision scar were demonstrated by radiologic, ultrasonographic, endoscopic and histologic methods by various authors.

Cesarean scar defect is a deficient uterine scar or scar dehiscence following a cesarean section involving myometrial discontinuity at the site of a previous cesarean section scar. Cesarean scar defects may be associated with many clinical problems such as ectopicpregnancy at the cesarean section scar, rupture of the uterus during a subsequent pregnancy, dysmenorrhea and abnormal uterine bleeding during the non-pregnant state. These complications are likely to be associated with poor uterine scar healing following cesarean sections.

Methods concerning closure of the uterine incision need to be considered with regards to benefit and potential harm in order to offer the best available surgical care to women undergoing cesarean section.

Sur-gical suturing technique and mechanical tension affecting the surgical wound are the most important factors related to the incisional integrity.

For this reason, investigators designed this prospective clinical study to analyze the effects of two different uterine suturing techniques. their aim was to compare the sparse closure of the uterine incision to classical one layer closure regarding short , mid and long term results. In deed, they compared :

* duration of surgery and calculated blood loss during surgery as short term results - incidence of postoperative defective healing of the uterine incision , thickness of the ultrasound imaged uterine scar as mid-term results .
* Incomplete uterine rupture, morbidly placental adhesion during subsequent pregnancy of these patients as long-term results.

DETAILED DESCRIPTION:
This is a secondary analyse of a first randomised trial comparing two caesarean techniques :

* Misgav Ladach with a one layer classic uterine closure.
* French ambulatory Caesarean section with a sparse uterine closure . The first trial is registred under the reference number : NCT03741907. 100 patients with an indication of an elective caesarean section were included in this trial : 50 had a one layer classic uterine closure and are enrolled in groupe 1 and 50 had a sparse uterine closure and are enrolled in groupe 2 .
* For the short term results investigators compared : duration of uterine sutures , visually estimated and calculated blood loss
* For the mid term results investigators are shuduling for all partient an hysterosonography 6 mounths after surgery and then will compare : incidence of postoperative defective healing of the uterine incision , thickness of the ultrasound imaged uterine scar as mid-term results .
* For the long term results investigators will interview patients 2 years after surgery in order to check for Incomplete uterine rupture, morbidly placental adhesion during subsequent pregnancy .

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* Cicatricial uterus with contraindication to vaginal delivery (uterus bi or multi-cicatricial, corporal uterine scar, intra-mural myomectomy, dystocic presentation)
* Fetal macrosomia with a weight greater than 4Kg
* Placenta previa

Exclusion Criteria:

* Patients who refuse to participate in the study
* prenatally diagnosed fetal pathology (intrauterine growth restriction, malformation, genetics disorders)
* adherent placenta, an adnexal mass or a myoma at the lower uterine segment
* Cesarean section in a context of medical or obstetrical emergency
* Caesarean section with a high risk of bleeding

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
uterine scar quality | 6 mounth after surgery
  ultrasound visualization of a defect on the internal wall of the uterine scar (niche)

SECONDARY OUTCOMES:
uterine scar thickness | 6 mounth after surgery
  ultrasound Measured thickness of the scar in sagittal and coronal section.
duration of surgery | during the caesarean section
  time spent for uterine closure
calculated blood loss | before and 24 hours after surgery
  post delivery hematocrit -predelivery hematocrit

CONTACTS AND LOCATIONS:
Locations (1):
- Kaouther Dimassi, Tunis, Sidi Daoued La Marsa, Tunisia

IPD SHARING:
Plan to Share IPD: No